CLINICAL TRIAL: NCT02600247
Title: Effects of Duloxetine on Pain Relief After Total Knee Arthroplasty in Central Sensitization Patient : A Randomized, Controlled, Double-Blind Trial
Brief Title: Effects of Duloxetine on Pain Relief After Total Knee Arthroplasty in Central Sensitization Patient
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The Catholic University of Korea (Other)
Responsible Party: Principal Investigator, Yong In, Proffesor, The Catholic University of Korea
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Duloxetine
Record Dates: First submitted 2015-11-05; First posted 2015-11-09 (Estimated); Last update posted 2015-11-09 (Estimated); Status verified 2015-11

CONDITIONS: Osteoarthritis
Keywords: Total knee arthroplasty; Duloxetine
MeSH Terms: conditions — Osteoarthritis | interventions — Duloxetine Hydrochloride; Celecoxib; Pregabalin; Acetaminophen; Tramadol; Oxycodone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Duloxetine group (Experimental): Experimental: Duloxetine group
  1. Phase I (preemptive): 1day before operation (30mg for 1 day)
  2. Phase II (maintenance): 6weeks after operation (30mg for 6 weeks) plus routine pain control (celecoxib, pregabalin, acetaminophen/tramadol, oxycodone)
  Other Name: cymbalta Drug: Celebrex, Lyrica, Ultracet, Ircodon
  Interventions: Drug: Duloxetine; Drug: celecoxib, Pregabalin, acetaminophen/tramadol, oxycodone
- routine pain control group (Active Comparator): Preemptive analgesia : celebrex 200mg 1C#1, Lyrica 150mg 1C#1 (preoperation. 2 hours), Patient controlled analgesia (postoperation 28 hours) During admission : celebrex 200mg#1, Ircodon 5mg 2T#2, Ultracet 2T#2 (Postoperation 1 week) Discharge medication: celebrex 200mg 1C#1 x 5Weeks, Ultracet 2T#2 x 1 week
  Other name : celecoxib, Pregabalin, acetaminophen/tramadol, oxycodone
  Interventions: Drug: celecoxib, Pregabalin, acetaminophen/tramadol, oxycodone

INTERVENTIONS:
Drug: Duloxetine — Experimental: Duloxetine group
  1. Phase I (preemptive): 1day before operation (30mg for 1 day)
  2. Phase II (maintenance): 6weeks after operation (30mg for 6 weeks) plus routine pain control (celecoxib, pregabalin, acetaminophen/tramadol, oxycodone)
  Other Name: cymbalta Drug: Celebrex, Lyrica, Ultracet, Ircodon
  Preemptive analgesia : celebrex 200mg 1C#1, Lyrica 150mg 1C#1 (preoperation. 2 hours), Patient controlled analgesia (postoperation 28 hours) During admission : celebrex 200mg#1, Ircodon 5mg 2T#2, Ultracet 2T#2 (Postoperation 1 week) Discharge medication: celebrex 200mg 1C#1 x 5Weeks, Ultracet 2T#2 x 1 week
  Other name : celecoxib, Pregabalin, acetaminophen/tramadol, oxycodone
  Arms: Duloxetine group
Drug: celecoxib, Pregabalin, acetaminophen/tramadol, oxycodone — Preemptive analgesia : celebrex 200mg 1C#1, Lyrica 150mg 1C#1 (preoperation. 2 hours), Patient controlled analgesia (postoperation 28 hours) During admission : celebrex 200mg#1, Ircodon 5mg 2T#2, Ultracet 2T#2 (Postoperation 1 week) Discharge medication: celebrex 200mg 1C#1 x 5Weeks, Ultracet 2T#2 x 1 week
  Other name : celecoxib, Pregabalin, acetaminophen/tramadol, oxycodone

SUMMARY:
This study aims to compare the effectiveness of duloxetine after total knee arthroplasty in Central sensitization patient. Central sensitization plays an important role in the chronic pain experienced by osteoarthritis patients.Elimination of the nociceptive input from the damaged joint by total joint arthroplasty was not always followed by a complete resolution of symptoms. Patients with high levels of preoperative pain and low pain thresholds had a higher risk of persistent pain after total knee arthroplasty (TKA), which has been interpreted as evidence of central sensitization. Thus, the presence of central sensitization before surgery in Osteoarthritis patients may be an important contributing factor to postoperative pain versus adequate analgesia. Preclinical models of central sensitization suggest that duloxetine is effective in the treatment of persistent pain. Investigators will compare the pain following TKA of central sensitization patients in duloxetine group (n=50) with those in non-duloxetine group (n=84). Investigators will classify the central sensitization patients by central sensitization inventory and divide the central sensitization patients in to 2 groups (duloxetine and non-duloxetine group) randomly. Investigators checks the visual assessment scale at preoperative, postoperative 1, 2,6,12 weeks. All participants will receive postoperative pain control after TKA using the same pain control regimen except duloxetine.

DETAILED DESCRIPTION:
Both groups of participants will receive pain control regimens as follows:

Preemptive analgesia : celebrex celecoxib, Lyrica Pregabalin, Patient controlled analgesia (postoperation 28 hours), During admission : celebrex 200mg#1, Ircodon 5mg 2Tablets#2, Ultracet 2T#2 (Postoperation 1 week) Discharge medication: celebrex 200mg 1Capsule#1 x 5 weeks, Ultracet 2T#2 x 1 week

Drug generic names: celecoxib (celebrex), Pregabalin (Lyrica), acetaminophen/tramadol (ultracet ER), oxycodone (Ircodon)

ELIGIBILITY:
Inclusion Criteria:

* Patients for total knee arthroplasty
* having medicare insurance
* CSI(Central sensitization inventory)> 40 (Central sensitization patient )

Exclusion Criteria:

* Rheumatoid arthritis
* Other inflammatory arthritis
* Neuropsychiatric patients
* Allergy or intolerance to study medications
* Patients with an ASA(American society of anesthesiologist) classification of IV (angina, congestive heart failure, dementia, cerebrovascular accident)
* Chronic gabapentin or pregabalin use (regular use for longer than 3 months)
* Chronic opioid use (taking opioids for longer than 3 months)
* Alcohol, drug abuser
* Narcotics addiction

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2015-11; Primary Completion 2016-11 (Estimated); Study Completion 2016-11 (Estimated)

PRIMARY OUTCOMES:
Visual pain scale | Preoperative & postoperative 1, 2, 6, 12 weeks

SECONDARY OUTCOMES:
SF(Short form)- 36 scale(Preoperative and postoperative 6, 12 weeks) | Preoperative and postoperative 6, 12 weeks
Brief pain inventory | Preoperative and postoperative 1, 6, 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Yong In, MD, PhD, Study Chair — Tthe Catholic Univerisity of Korea Seoul St Mary's hospital